CLINICAL TRIAL: NCT06342830
Title: Comparison of the Effects of Different Natural and Synthetic Intracanal Medicaments on the Healing of Periapical Lesion in Retreatment Cases (A Randomized Clinical Trial)
Brief Title: Comparing the Effect of Different Intracanal Dressing on Failed Root Canal Treated Cases on Periapical Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rawda Baghdady, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: End 20-05 P
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Periapical Disease
MeSH Terms: conditions — Periapical Diseases | interventions — Ciprofloxacin; Ibuprofen; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nanocurcumin gel . (Experimental): Preparation Method: Olive oil (5%), surfactant (Tween 80 (8%)) and co-surfactant (PEG 400 (2%)) were used as excipients and their selection was based on the solubility of curcumin. A high-energy ultrasonication techniquewas used to prepare the Cur-NE. Curcumin (0.3%) was dissolved in oil /surfactant/ co-surfactant mixture and stirred till obtaining clear solution. The mixture was microtitrated with distilled water (85 %) to achieve a coarse emulsion. A 20 kHz ultrasonic processor was used for the production of the desired nano-emulsion.
  Gel Preparation:
  0.4gm of Carboxymethyl cellulose (Loba CHIME, india) was sprinkled gently and gradually over the solution of Cur NE 0.3% under mild temperature with vigorous stirring to get homogenous gel
  Interventions: Drug: nanocurcumin gel
- Curcumin gel (Experimental): curcumin 250 mg powder + carboxymethyl cellulose 300mg+distilled water to 10ml
  Interventions: Drug: Curcumin Gel
- Ciprofloxacin 500 mg +Ibuprofen 400 mg (Experimental): Ciprofloxacin 500 mg +ibuprofen 400mg powder +carboxymethyl cellulose 300 mg +distilled water to 10 ml
  Interventions: Drug: Ciprofloxacin 500 mg +ibuprofen 400mg
- calcium hydroxide (Active Comparator): Metapaste
  Interventions: Drug: Metapaste [calcium hydroxide paste (control group)]

INTERVENTIONS:
Drug: nanocurcumin gel — firstly patient anesthetized, rubber dam isolation , disinfect the crown with 10%H2O2, saline then sodium hypochlorite solution 2.5% then 5% sodium thiosulphate solution to inhibit the effect of NaOHCl then removal of old coronal restoration, disinfection of pulp chamber by the same previous protocol removal of old root canal filling with gates glidden drills and H files , taken first sample S1 from canal with paper point after using saline wash and scrubbing the canal wall the paper points left for 1 min in the canal then preparation of canal with edge endo files till size 45 taper 0.4 and NaOHCL 2.5% between each file and the next finally 5% sodium thiosulphate to inhibit the antibacterial effect of sodium hypochlorite irrigation then saline irrigation and scrubbing the canal wall and placement of paper points for 1min to taken second sample S2, then dryness of canal and placement of nanocurcumin gel until shown fill the canal under magnification and by using lentulospirals
  Arms: Nanocurcumin gel .
Drug: Curcumin Gel — firstly patient anesthetized, rubber dam isolation , disinfect the crown with 10%H2O2, saline then sodium hypochlorite solution 2.5% then 5% sodium thiosulphate solution to inhibit the effect of NaOHCl then removal of old coronal restoration, disinfection of pulp chamber by the same previous protocol removal of old root canal filling with gates glidden drills and H files , taken first sample S1 from canal with paper point after using saline wash and scrubbing the canal wall the paper points left for 1 min in the canal then preparation of canal with edge endo files till size 45 taper 0.4 and NaOHCL 2.5% between each file and the next finally 5% sodium thiosulphate to inhibit the antibacterial effect of sodium hypochlorite irrigation then saline irrigation and scrubbing the canal wall and placement of paper points for 1min to taken second sample S2, then dryness of canal and placement of curcumin gel until shown fill the canal under magnification and by using lentulospirals
  Arms: Curcumin gel
Drug: Ciprofloxacin 500 mg +ibuprofen 400mg — firstly patient anesthetized, rubber dam isolation , disinfect the crown with 10%H2O2, saline then sodium hypochlorite solution 2.5% then 5% sodium thiosulphate solution to inhibit the effect of NaOHCl then removal of old coronal restoration, disinfection of pulp chamber by the same previous protocol removal of old root canal filling with gates glidden drills and H files , taken first sample S1 from canal with paper point after using saline wash and scrubbing the canal wall the paper points left for 1 min in the canal then preparation of canal with edge endo files till size 45 taper 0.4 and NaOHCL 2.5 % between each file and the next finally 5% sodium thiosulphate to inhibit the antibacterial effect of sodium hypochlorite irrigation then saline irrigation and scrubbing the canal wall and placement of paper points for 1min to taken second sample S2, then dryness of canal and placement of ciprofloxacin + ibuprofen gel until fill the canal under magnification and by using lentulospirals
  Arms: Ciprofloxacin 500 mg +Ibuprofen 400 mg
Drug: Metapaste [calcium hydroxide paste (control group)] — firstly patient anesthetized, rubber dam isolation , disinfect the crown with 10%H2O2, saline then sodium hypochlorite solution 2.5% then 5% sodium thiosulphate solution to inhibit the effect of NaOHCl then removal of old coronal restoration, disinfection of pulp chamber by the same previous protocol removal of old root canal filling with gates glidden drills and H files , taken first sample S1 from canal with paper point after using saline wash and scrubbing the canal wall the paper points left for 1 min in the canal then preparation of canal with edge endo files till size 45 taper 0.4 and NaOHCL 2.5 % between each file and the next finally 5% sodium thiosulphate to inhibit the antibacterial effect of sodium hypochlorite irrigation then saline irrigation and scrubbing the canal wall and placement of paper points for 1min to taken second sample S2, then dryness of canal and placement of calcium hydroxide paste until fill the canal under magnification by using lentulospirals
  Arms: calcium hydroxide

SUMMARY:
The goal of this clinical trial is to compare the effects of different intracanal medication between endodontic retreatment visits in previously failed root canal treatment patients (single root canal anteriors or premolars teeth). The main question it aims to answer are:

* Is natural and synthetic intracanal Medicament effective in reducing or complete healing of Periapical lesions or not? the researchers will compare the effect of different intracanal dressing including:
* nanocurcumin gel
* curcumin gel
* ciprofloxacin +ibuprofen gel
* calcium hydroxide Paste as control group in between the endodontic retreatment visits to see if these medicaments work well on periapical lesion healing this outcome measured by Cone beam CT at base and after 1 year follow up period

ELIGIBILITY:
Inclusion Criteria:

* Medically free Patients
* both sex includes male and females
* Patients age between 20-60
* Patients agreement positively to share in the study
* patient able to sign informed consent
* on clinical and radiographic examinations, the included teeth maxillary and mandibular single root canal anteriors or premolars suffering from failed endodontic treatment with periapical lesion

Exclusion Criteria:

* badly broken down teeth indicated for extraction or with difficult isolation
* teeth with former procedural errors as ledge, perforation or instrument separation
* Medically compromised patients
* patients with history of receiving antibiotics within a month before starting study
* periodontally affected teeth by pocket depth & > 4mm

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
healing of periapical lesion | 1 year
  measured radiographically the periapical lesion volmetric changes by CBCT between preoperative and after1 year follow up

SECONDARY OUTCOMES:
antibacterial effect (CFU) | at first visit : S1 :baseline sample, S2 : sample immediately after chemomechanical procedure , at second visit S3: sample after 7 days of placement medication
  Three samples S1 after removal of old root canal filling , S2 after mechanical Preparation , S3 after 7 days of placement of intracanal dressing measuring total bacterial count by colony forming unit each sample cultured and incubated for 24hours and bacterial counting measured
Interappointment Pain | 6,12, 24, 48, 72 hours after 1st visit
  measured by Numerical Rating Scale (NRS) which is an 11-point scale consisting of numbers from 0 through 10 0 reading represents "no pain"
  1- 3 readings represent "mild pain" 4- 6 readings represent "moderate pain" 7- 10 readings represent "severe pain" No or mild pain was considered as success while moderate or severe pain were regarded as failure.

CONTACTS AND LOCATIONS:
Overall Officials: Rawda MO Baghdady, Principal Investigator — faculty of dentistry, zagazig university; sarah H Fahmy, Study Chair — faculty of dentistry, Ain Shams university; karim M El Batouty, Study Director — faculty of dentistry, Ain Shams university
Locations (1):
- faculty of dentistry, Ain shams university, Cairo, Egypt

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT06342830/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT06342830/ICF_001.pdf